CLINICAL TRIAL: NCT03238846
Title: Outcomes of Differentiated Models of Care: Multi-Month Dispensing (MMD) and Community ART Refill Groups (CARGs) in Stable ART Patients
Brief Title: Operations Research of the 'Real World' Effectiveness of Multi-Month Dispensing of ART for Stable Patients in CARGs in Zimbabwe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kheth'Impilo (Other)
Collaborators: Ministry of Health and Child Welfare, Zimbabwe (Other); EQUIP Innovation for Health (Unknown); Organization for Public Health Interventions and Development (OPHID) (Unknown); Family Health International (FHI 360) (Unknown); Population Services International (PSI) (Unknown)
Responsible Party: Principal Investigator, Dr Nicoletta Mabhena, EQUIP Technical Lead, Kheth'Impilo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MMSD Study; MRCZ/A/2168 (Other: MRCZ)
Record Dates: First submitted 2017-07-27; First posted 2017-08-03 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: A prospective, parallel, cluster randomized noninferiority trial with three study arms will be conducted. In this study, a health facility is a cluster or site. Study sites were purposively selected from Chitungwiza Municipality, Masvingo Provincial districts, Matebeleland South Provincial districts, and Mberengwa district where USAID partners are currently implementing CARGs. Thirty clusters were selected and randomized in two strata per geographic location (urban and rural) to the three study arms. Outcomes will be assessed after 12 and 24 months,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3MF: 3-month ART dispensing at facilities (No Intervention): Ten sites at which patients will receive standard of care where ART is dispensed three monthly from the facility based on usual practice at the clinic. The approach will be consistent with applicable country guidelines at the time of study.
- 3MC: 3-month ART dispensing in CARGs (Experimental): Ten sites at which patients will receive ART dispensed three monthly in CARGs. Providers at facilities will assist in the formation of CARGs and will provide all enrolled patients with a 3 month supply of ART and associated HIV medications. All other aspects of care will be as per standard of care for the enrolling clinic.
  Interventions: Other: Three month dispensing of ART in CARGs
- 6MC: 6-month ART dispensing in CARGs (Experimental): Ten sites at which patients will receive ART dispensed six monthly in CARGs. Providers at facilities will assist in the formation of CARGs and will provide all enrolled patients with a 6 month supply of ART and associated HIV medications. All other aspects of care will be as per standard of care for the enrolling clinic.
  Interventions: Other: Six month dispensing of ART in CARGs

INTERVENTIONS:
Other: Three month dispensing of ART in CARGs — Patients enrolled in the three-month ART dispensing arm will receive a 90-day supply of ART in CARGs from their provider for the duration of the study. Each CARG will consist of 6-12 stable patients on ART and will meet in the community and select a group member to collect their ART at the facility every 3 months. Patients can have unscheduled clinic visits when unwell. Viral loads for the group will be collected at 12 and 24 months at the facility.
  Arms: 3MC: 3-month ART dispensing in CARGs
Other: Six month dispensing of ART in CARGs — Patients enrolled in the three-month ART dispensing arm will receive a 90-day supply of ART in CARGs from their provider for the duration of the study. Each CARG will consist of 6-12 stable patients on ART and will meet in the community and select a group member to collect their ART at the facility every 6 months. Patients can have unscheduled clinic visits when unwell. Viral loads for the group will be collected at 12 and 24 months at the facility.
  Arms: 6MC: 6-month ART dispensing in CARGs

SUMMARY:
This study aims to evaluate the effectiveness of two strategies for multi-month dispensing (MMD) of ART in Community ART Refill Groups (CARGs) on retention, virologic suppression, and cost compared to standard of care.

This study is a three-arm cluster-randomized controlled trial conducted among 5,760 stable HIV-positive patients) in Zimbabwe to compare outcomes of three antiretroviral therapy (ART) dispensing models. Outcomes of retention in care, virologic suppression, and cost effectiveness will be investigated in 30 purposively selected clusters (facilities) which are randomized into three arms; standard of care (3 months dispensing at facilities), three-month dispensing in CARGs, and six-month dispensing in CARGs. Each study arm will have 10 clusters stratified into 2 urban and 8 rural. Study participants will be followed, and outcomes will be measured at 12 months and 24 months. Qualitative research will be conducted at baseline, 12 months, and 24 months (20 participant Focus Group Discussion (FGDs) and 20 provider Key Informant Interview (KII) at each interval) to understand patient and health provider acceptability of multi-month dispensing of ART within CARGs. Other outcomes of interest include measuring gains of facility decongestion and feasibility of multi-month dispensing of ART within CARGs. Cost analysis will include comparisons of patient level costs, cost per patient outcomes and cost effectiveness across the three study arms.

DETAILED DESCRIPTION:
This study will use a cluster (facility) randomized trial with 3 arms; patients receiving 3 monthly ART supply at facilities-standard of care (3MF) (Control group), patients receiving 3 monthly ART supply at newly formed CARGs (3MC) and patients receiving 6 monthly ART supply at newly formed CARGs (6MC). Participants will be followed up for 24 months. A total of 30 study clusters (facilities) will be randomization, into the three study arms; 10 clusters per arm stratified 2 urban, 8 rural.

Study Setting and study population The study population is HIV-infected adults over the age of 18 years recruited from health facilities in U.S. President's Emergency Plan for AIDS Relief (PEPFAR) Zimbabwe scale-up districts (using existing national records of patients in the ART registers) that have been stable on a standard first-line ART treatment regimen for at least 6 months.

Facilities from Chitungwiza Municipality, Matebeleland South Province, Masvingo Province and Mberengwa district will be purposively selected to be the urban/periurban and rural settings in the study. These areas were selected as they have PEPFAR Zimbabwe scale-up priority facilities, high numbers of patients on ART and have prioritized implementation of CARGs. These locations are also viewed to be good representations of PEPFAR Zimbabwe scale-up priority facilities, hence are likely to improve the generalizability of the study findings to the study population. As contexts differ between rural and urban/periurban settings, it is important to determine the effectiveness of MMD within CARGs within both contexts.

Sampling and Sample size Sample sizes were determined for a cluster-randomized noninferiority trial, using PASS v.14 (TM) software. Sample size estimates were calculated for the primary outcome of retention in care at 12 months. The probability of patient attrition twelve months after study enrolment in the control group (3MF) is assumed to be 5%, derived from the relative difference in patient retention between 12 and 24 months from the 2015 Zimbabwe UNAIDS Global AIDS Response progress report. An intracluster correlation coefficient (ICC) of 0.01 for patient retention/attrition amongst stable ART patients is assumed. The noninferiority limit is specified as 3.25%. Assuming α=0.05, power of 85%, using one-sided Z-test (unpooled) test statistic, 182 participants per facility will be required with a total sample size of 5460 participants. A sample size re-estimation during accrual will increase the total sample size to approximately 5760; 192 enrolled participants per study site and 1,920 participants per arm. As retention in care is the primary outcome, no adjustment for loss to follow-up needs to be made.

Study procedures As this is operational research, the study will not interfere with routine patient management and will follow national guidelines. The health care worker assesses each patient's clinical notes to establish stability and study inclusion. Once informed consent is obtained, a baseline questionnaire will be applied to record demographic characteristics and the patients clinical and ART history. Patients will receive care based on their study ARM and relevant SOP. Patient files and CARG tools will be reviewed and data collected at each ART refill. Viral loads will be repeated annually.

Data Collection The study will use both qualitative and quantitative methods. The data sources will include patient clinic notes, electronic patient management system (ePMS), CARG monitoring data collection tools. In addition, variables to control for confounding in the analysis for outcomes of interest will be collected at baseline through a short cross-sectional survey. A pre-and-24-month post survey time-flow evaluation of patient waiting times to assess gains of facility decongestion will be conducted. Feasibility of MMD of ART within CARGs will be measured prospectively at baseline, 12 and 24 months. To understand the acceptability of CARGs by patients and service providers; patient satisfaction, and improvement in quality of care at the facilities, 20 patient FGDs and 20 heath care provider KII will be conducted at baseline, 12 and 24 months. A micro-costing approach supplemented by a macro-costing approach of fixed costs will be utilized to measure cost outcomes. A resource use form will collect information per patient through retrospective review of clinic records. Start up costs will be included under each arm. Data to assess patient level costs will be collected from a randomly selected sub-sample of 365 patients per arm at baseline, 12 months and 24 months.

Data analysis Quantitative data will be analyzed using STATA 14. An intention-to-treat analysis will be performed for the primary outcome of retention in care, in which all patients and clinics will be analyzed in the group to which they were originally assigned. Risk differences between arms will be compared with binomial population averaged generalized estimating equations using an identity link and an exchangeable correlation matrix, specifying for clustering by facility. Viral load suppression analyzed using log-binomial regression, generalized estimating equations will be used to estimate risk ratios between the study arms, specifying for clustering by facility and using an exchangeable correlation matrix. Average patient waiting times will be compared between study arms using linear regression.

Content qualitative analysis will be conducted using Atlas Ti, A cost outcomes analysis will be conducted from the provider perspective. Average cost per yield rates (cost per client retained in care, cost per client virally suppressed, cost per patient per year) will be calculated. An incremental cost-effectiveness ratio (ICER) for the will be calculated; ICER threshold comparison as recommended by World Health Organisation (WHO) will be employed. Average patient costs will be from the patient's perspective. Startup costs for each service delivery model will also be analyzed.

RISKS / BENEFITS TO PARTICIPANTS There may be no direct benefit to participants who take part in this study, beyond benefits related to their routine ART medication that would have been achieved otherwise. Information learned in this study may be of benefit to participants and others in the future, particularly information that may lead to optimized treatment guidelines for HIV-infected stable patients on ART.

As this is operational research, study procedures are routine clinical care associated with minimal risk to participants. All patients will attend routine clinic visits to be assessed for new Opportunistic infections (OIs), pregnancy, drug-drug interactions or side effects of medications. This will ensure that patients who develop co-morbidities or become pregnant during the study receive standard care, although they will not be excluded from the study.

REIMBURSEMENTS AND COMPENSATION As participants of FGDs may use transport money to the discussion venue, this will be reimbursed. Those who are part of a FGD will receive snacks after the discussion. CARGs will receive a bag to carry drugs from the clinic back to their communities. This will be made clear to all study participants during the informed consent process.

CONFIDENTIALITY ASSURANCES Participant information will not be released without written permission to do so except as necessary for review, monitoring, and/or auditing. All study-related information will be stored securely. Participant research records will be stored in locked areas with access limited to study staff. case record files (CRFs), and other documents that may be transmitted off-site will be identified by patient identifier only. Likewise, communications between study staff and the investigators regarding individual participants will identify participants by patient identifier only. The patient identifier will be an anonymized key to identify unique subjects and will be used for data pooling, transfer, storage, manipulation and analysis. Personal identifying data will not be available to the investigators. Study sites will store study records that bear participant names or other personal identifiers separately from records identified by patient identifier. Lists, logbooks, appointment books, and any other documents that link the patient identifier to personal identifying information at the facilities should be stored in a separate, locked location in an area with limited access. Electronic data will be stored on password secured servers, which will be backed-up on a regular basis. Data will be presented in aggregate form only.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and willing and able to provide written informed consent for participation in this study
* Willing to be part of a CARG if in a facility that has been randomized to 3MC or 6MC,
* Confirmed HIV-1 infection based on the Zimbabwe National HIV testing algorithm.
* On ART ≥ 6 months
* On first line ART regimen
* No drug toxicity/tolerability issues within the prior 6 months
* No active opportunistic infection suspected (including TB) and not treated for an opportunistic infection in the last 30 days
* Viral load < 1000 copies/ml done at baseline of the study
* Weight ≥ 35kgs

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* On alternative first line or second line regimen
* ARV toxicity or tolerability issue within the prior 6 months
* Co-morbidities requiring facility visits more often than 3 months if in the 3MC/3MF ARMS and 6 monthly if in the 6MC ARM
* Viral load > lower limit of standard assay (>1000) within the prior 6 months
* Confirmed pregnancy, or less than 18 months postpartum.
* Weight criteria is less than 35kgs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4676 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Retention in care | 12 months
  To determine if stable ART patients receiving 3 monthly dispensing of ART within CARGs have noninferior retention in care than stable ART patients receiving 3 monthly dispensing at health facilities after 12 months.
Retention in care | 12 months
  To determine if stable ART patients receiving 6 monthly dispensing of ART within CARGs have noninferior retention in care than stable ART patients receiving 3 monthly dispensing at health facilities after 12 months.
Measure change in retention in care | 12 and 24 months
  To determine if stable ART patients within CARGs receiving 6 monthly dispensing of ART have noninferior retention in care than stable ART patients receiving 3 monthly dispensing within CARGs after 12 months

SECONDARY OUTCOMES:
Virologic suppression | 12 months
  To determine if stable ART patients receiving 3 and 6 monthly dispensing of ART within CARGs have noninferior viral suppression than stable ART patients receiving 3 monthly dispensing at health facilities after 12 months.
Measure change in virologic suppression | 12 and 24 months
  To determine if stable ART patients within CARGs receiving 6 monthly dispensing have noninferior viral suppression than stable ART patients receiving 3 monthly dispensing within CARGs after 12 months and 24 months.
Measure cost effectiveness at 2 time points | 12 and 24 months
  To determine the cost-effectiveness of dispensing of ART for three and six months within CARGs compared to three months in facilities (standard of care). Cost-effectiveness will be estimated as the average cost per successful outcome (patient retained at 12 and 24 months)
Measure change in patient level benefits of implementing CARGs | 12 and 24 months
  To determine patient-level benefits of implementing CARGs with 3 monthly and 6 monthly dispensing (effects on cost of accessing care, productivity benefits and informal care effects).
Measuring change in feasibility of multi-month dispensing of ART within CARGs | 12 and 24 months
  To determine the feasibility of the introduction of multi-month dispensing of ART within CARGs and distribution in Zimbabwe (policy, supply chain management, and implementation).
Measure change in acceptability of CARGs | 12 and 24 months
  To determine the acceptability of 3 and 6 monthly dispensing of ART within CARGs by patients and service providers.
Measuring change in gains of facility decongestion | 12 and 24 months
  To assess if there are any measurable gains made by decongesting facilities following the introduction of multi-month dispensing of ART within CARGs.

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Ngorima-Mabhena, MBChB, MSc Epidemiology, Principal Investigator — Kheth'Impilo
Locations (30):
- Zimbabwe (30):
  - Seke North Clinic, Chitungwiza, Harare
  - Seke South Clinic, Chitungwiza, Harare
  - St Mary's Clinic, Chitungwiza, Harare
  - Zengeza Clinic, Chitungwiza, Harare
  - Chimombe Rural Hospital, Gutu, Masvingo Province
  - Chinyika Rural Hospital, Gutu, Masvingo Province
  - Gutu Mission Hospital, Gutu, Masvingo Province
  - Gutu Rural Hospital, Gutu, Masvingo Province
  - Bota Rural Hospital, Zaka, Masvingo Province
  - Bvukururu Clinic, Zaka, Masvingo Province
  - Chiredzana Clinic, Zaka, Masvingo Province
  - Harava Rural Health Centre, Zaka, Masvingo Province
  - Siyawareva Clinic, Zaka, Masvingo Province
  - Beitbridge Hospital, Beitbridge, Matebeleland South
  - Chamnangana, Beitbridge, Matebeleland South
  - Chaswingo, Beitbridge, Matebeleland South
  - Dulibadzimu, Beitbridge, Matebeleland South
  - Makakabule, Beitbridge, Matebeleland South
  - Shabwe, Beitbridge, Matebeleland South
  - Chidembeko Mission Hospital, Mberengwa, Midlands Province
  - Jeka Mission Hospital, Mberengwa, Midlands Province
  - Masase Mission Hospital, Mberengwa, Midlands Province
  - Mataga RHC, Mberengwa, Midlands Province
  - Mberengwa Hospital, Mberengwa, Midlands Province
  - Mnene Mission Hospital, Mberengwa, Midlands Province
  - Mposi Mission Hospital, Mberengwa, Midlands Province
  - Musume Mission Hospital, Mberengwa, Midlands Province
  - Mwanezi RHC, Mberengwa, Midlands Province
  - Negove Clinic, Mberengwa, Midlands Province
  - Svuure Clinic, Zaka, Midlands Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fatti G, Ngorima-Mabhena N, Tiam A, Tukei BB, Kasu T, Muzenda T, Maile K, Lombard C, Chasela C, Grimwood A. Community-based differentiated service delivery models incorporating multi-month dispensing of antiretroviral treatment for newly stable people living with HIV receiving single annual clinical visits: a pooled analysis of two cluster-randomized trials in southern Africa. J Int AIDS Soc. 2021 Oct;24 Suppl 6(Suppl 6):e25819. doi: 10.1002/jia2.25819. PMID 34713614
- [Derived] Lopes J, Grimwood A, Ngorima-Mabhena N, Tiam A, Tukei BB, Kasu T, Mahachi N, Mothibi E, Tukei V, Chasela C, Lombard C, Fatti G. Out-of-Facility Multimonth Dispensing of Antiretroviral Treatment: A Pooled Analysis Using Individual Patient Data From Cluster-Randomized Trials in Southern Africa. J Acquir Immune Defic Syndr. 2021 Dec 15;88(5):477-486. doi: 10.1097/QAI.0000000000002797. PMID 34506343
- [Derived] Fatti G, Ngorima-Mabhena N, Mothibi E, Muzenda T, Choto R, Kasu T, Tafuma TA, Mahachi N, Takarinda KC, Apollo T, Mugurungi O, Chasela C, Hoffman RM, Grimwood A. Outcomes of Three- Versus Six-Monthly Dispensing of Antiretroviral Treatment (ART) for Stable HIV Patients in Community ART Refill Groups: A Cluster-Randomized Trial in Zimbabwe. J Acquir Immune Defic Syndr. 2020 Jun 1;84(2):162-172. doi: 10.1097/QAI.0000000000002333. PMID 32097252
- [Derived] Fatti G, Ngorima-Mabhena N, Chirowa F, Chirwa B, Takarinda K, Tafuma TA, Mahachi N, Chikodzore R, Nyadundu S, Ajayi CA, Mutasa-Apollo T, Mugurungi O, Mothibi E, Hoffman RM, Grimwood A. The effectiveness and cost-effectiveness of 3- vs. 6-monthly dispensing of antiretroviral treatment (ART) for stable HIV patients in community ART-refill groups in Zimbabwe: study protocol for a pragmatic, cluster-randomized trial. Trials. 2018 Jan 29;19(1):79. doi: 10.1186/s13063-018-2469-y. PMID 29378662